CLINICAL TRIAL: NCT05554900
Title: The Efficacy, Safety and Prognosis of Preventive Regenerative Peripheral Nerve Interface(RPNI) Reconstruction in Amputees: Study Protocol for a Cohort Study
Brief Title: The Efficacy of Preventive Regenerative Peripheral Nerve Interface(RPNI) Reconstruction in Amputees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Li Guangxue, Deputy Chief Physician, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: lgx2022
Record Dates: First submitted 2022-09-03; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Amputation Neuroma
Keywords: Amputation; Regenerative peripheral nerve interface; Neuroma
MeSH Terms: conditions — Neuroma

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The investigator who perform the operations cannot be blinded because of the use of manual techniques.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (No Intervention): The control group received traditional amputation.The proximal nerve is blocked with lidocaine and cut off. The end of the nerve retracted as far as possible and the bleeding point is ligated if necessary.
- The experimental group（RPNIs group） (Experimental): The experimental group received regenerative peripheral nerve interface（RPNI） surgery.
  Interventions: Procedure: preventive regenerative peripheral nerve interface reconstruction

INTERVENTIONS:
Procedure: preventive regenerative peripheral nerve interface reconstruction — Each RPNI unit consists of nerve stump and free autologous muscle graft that is cut off from healthy muscle of the amputated limb. The muscle graft is approximately 30×15×5 mm.The ends of the transected nerve are placed within the muscle belly of the free muscle grafts in an orientation that is parallel to the muscle fibers. Next, the nerve is secured distally with 6-0 non-absorbable monofilament sutures in an epimysial-to-epineurial fashion. The nerve is then wrapped around completely via muscle graft and epimysial securing sutures. All RPNI units are placed in areas remote from the surgical incision and from the weight-bearing surface of the limb.
  Arms: The experimental group（RPNIs group）

SUMMARY:
The trial will be carried out in Peking University People's Hospital. The whole trial will last 3 years. Amputees from orthopedics and vascular surgery will be distributed into two groups randomly and receive different treatments including traditional resection and regenerative peripheral nerve interface(RPNI) surgery.The pain outcome,the impact of post-amputation pain on life and the utilization rate of prostheses will be collected to study the efficacy, safety and prognosis of preventive regenerative peripheral nerve interface reconstruction in amputees.

Investigators believe that RPNI can effectively reduce the incidence of post-amputation pain, reduce the degree of pain, improve the wearing rate of prostheses, and help patients return to normal life.

ELIGIBILITY:
Inclusion Criteria:

* Perform traditional amputation and nerve disconnection or RPNIs in Peking University People's Hospital
* Age≥6 years
* Follow-up time≥12 weeks

Exclusion Criteria:

* Follow-up time<12 weeks
* Age<6 years
* Preoperative complications included cervical spondylosis, lumbar spinal stenosis, piriformis syndrome, cubital tunnel syndrome and other peripheral nerve entrapment syndrome

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
postamputation pain | 12 weeks at least after surgery
  Patient-Reported Outcomes Measurement Information System (NRS, PROMIS) were used to assess postamputation pain.The intensity of pain is described by 11 points from 0 (painless) to 10 (the most severe pain).

SECONDARY OUTCOMES:
Prosthesis wearing | 12 weeks at least after surgery
  Whether the subject wears a prosthetic limb, and if so, what kind of prosthetic limb is worn.
Tumor recurrence and metastasis | 12 weeks at least after surgery
  Whether there is tumor recurrence or metastasis.
Quality of life | 12 weeks at least after surgery
  The medical outcomes study-short from(MOS-SF 36) is used to evaluate the difference between the RPNIs group and the control group in the quality of life after amputation.The SF-36 scale consists of 36 questions with eight dimensions:physiological function, role-physiological, physical pain, general health, vitality, social function, role-emotional, and mental health. The scoring method was used for each dimension, ranging from 0 to 100 points. The higher the score, the better the health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watson J, Gonzalez M, Romero A, Kerns J. Neuromas of the hand and upper extremity. J Hand Surg Am. 2010 Mar;35(3):499-510. doi: 10.1016/j.jhsa.2009.12.019. PMID 20193866
- [Background] Zimmermann M. Pathobiology of neuropathic pain. Eur J Pharmacol. 2001 Oct 19;429(1-3):23-37. doi: 10.1016/s0014-2999(01)01303-6. PMID 11698024
- [Background] Bowsher D. Human "autotomy". Pain. 2002 Jan;95(1-2):187-9. doi: 10.1016/s0304-3959(01)00389-x. PMID 11790481
- [Background] Niederberger E, Kuhlein H, Geisslinger G. Update on the pathobiology of neuropathic pain. Expert Rev Proteomics. 2008 Dec;5(6):799-818. doi: 10.1586/14789450.5.6.799. PMID 19086860
- [Background] McFarland LV, Hubbard Winkler SL, Heinemann AW, Jones M, Esquenazi A. Unilateral upper-limb loss: satisfaction and prosthetic-device use in veterans and servicemembers from Vietnam and OIF/OEF conflicts. J Rehabil Res Dev. 2010;47(4):299-316. doi: 10.1682/jrrd.2009.03.0027. PMID 20803400
- [Background] Davis RW. Phantom sensation, phantom pain, and stump pain. Arch Phys Med Rehabil. 1993 Jan;74(1):79-91. PMID 8380543
- [Background] Vlot MA, Wilkens SC, Chen NC, Eberlin KR. Symptomatic Neuroma Following Initial Amputation for Traumatic Digital Amputation. J Hand Surg Am. 2018 Jan;43(1):86.e1-86.e8. doi: 10.1016/j.jhsa.2017.08.021. Epub 2017 Sep 23. PMID 28951100
- [Background] Ives GC, Kung TA, Nghiem BT, Ursu DC, Brown DL, Cederna PS, Kemp SWP. Current State of the Surgical Treatment of Terminal Neuromas. Neurosurgery. 2018 Sep 1;83(3):354-364. doi: 10.1093/neuros/nyx500. PMID 29053875
- [Background] Poppler LH, Parikh RP, Bichanich MJ, Rebehn K, Bettlach CR, Mackinnon SE, Moore AM. Surgical interventions for the treatment of painful neuroma: a comparative meta-analysis. Pain. 2018 Feb;159(2):214-223. doi: 10.1097/j.pain.0000000000001101. PMID 29189515
- [Background] Barbour JR, Yee A, Moore AM, Trulock EP, Buchowski JM, Mackinnon SE. Cadaveric nerve allotransplantation in the treatment of persistent thoracic neuralgia. Ann Thorac Surg. 2015 Apr;99(4):1414-7. doi: 10.1016/j.athoracsur.2014.06.092. PMID 25841822
- [Background] Elliot D. Surgical management of painful peripheral nerves. Clin Plast Surg. 2014 Jul;41(3):589-613. doi: 10.1016/j.cps.2014.03.004. PMID 24996473
- [Background] Lipinski LJ, Spinner RJ. Neurolysis, neurectomy, and nerve repair/reconstruction for chronic pain. Neurosurg Clin N Am. 2014 Oct;25(4):777-87. doi: 10.1016/j.nec.2014.07.002. Epub 2014 Aug 14. PMID 25240664
- [Background] Kuiken TA, Miller LA, Lipschutz RD, Lock BA, Stubblefield K, Marasco PD, Zhou P, Dumanian GA. Targeted reinnervation for enhanced prosthetic arm function in a woman with a proximal amputation: a case study. Lancet. 2007 Feb 3;369(9559):371-80. doi: 10.1016/S0140-6736(07)60193-7. PMID 17276777
- [Background] Peters BR, Russo SA, West JM, Moore AM, Schulz SA. Targeted muscle reinnervation for the management of pain in the setting of major limb amputation. SAGE Open Med. 2020 Sep 15;8:2050312120959180. doi: 10.1177/2050312120959180. eCollection 2020. PMID 32974021
- [Background] Santosa KB, Oliver JD, Cederna PS, Kung TA. Regenerative Peripheral Nerve Interfaces for Prevention and Management of Neuromas. Clin Plast Surg. 2020 Apr;47(2):311-321. doi: 10.1016/j.cps.2020.01.004. Epub 2020 Feb 1. PMID 32115057
- [Background] Kubiak CA, Kemp SWP, Cederna PS, Kung TA. Prophylactic Regenerative Peripheral Nerve Interfaces to Prevent Postamputation Pain. Plast Reconstr Surg. 2019 Sep;144(3):421e-430e. doi: 10.1097/PRS.0000000000005922. PMID 31461024
- [Background] Woo SL, Urbanchek MG, Cederna PS, Langhals NB. Revisiting nonvascularized partial muscle grafts: a novel use for prosthetic control. Plast Reconstr Surg. 2014 Aug;134(2):344e-346e. doi: 10.1097/PRS.0000000000000317. No abstract available. PMID 25068369